CLINICAL TRIAL: NCT03153670
Title: 3T MRI in Patients With Deep Brain Stimulation (DBS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Andres M. Lozano, Neurosurgeon, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-8255
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Neuro-Degenerative Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- fMRI-based programming (Experimental): DBS patients will undergo fMRI scanning while on different stimulation settings. The results will be fed to the programming clinician (movement disorder neurologist) to aid the conventional programming process at the clinician's discretion.
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — DBS patients will undergo fMRI scanning. For each patient, scans will be performed using a selection of DBS settings. fMRI responses will be analysed to evaluate brain responses on different DBS settings. These results will be provided to the programming clinician to guide them choose the optimal setting for each patient at the clinician's discretion.

SUMMARY:
Deep brain stimulation (DBS) is an established treatment for advanced Parkinson's disease, medically refractory tremor, dystonia and obsessive compulsive disorder. Several hypotheses driven DBS trials are underway to study modulation of circuit dysfunction in other neurological and psychiatric disorders like epilepsy, Alzheimer's disease and depression. Recent reports suggest profound effects of DBS on the anatomy and function of downstream areas in the brain. For example electrical stimulation of limbic circuits is associated with increase in hippocampal neurogenesis. Similarly, stimulation of subthalamic nucleus (STN) or globus pallidus (GPi) results in activation of cortical motor circuits. Non-invasive imaging modalities are increasingly being employed in these investigations to better understand the effects of DBS on the structure and function of the brain.

There have been important advances in MRI and we now have MRI which provides higher resolution and higher quality brain images. More specifically, the investigators propose to use MRI to perform functional magnetic resonance imaging (i.e. fMRI) to assess the effects of deep brain stimulation on brain function and to assess whether fMRI can be used as an adjunct to improve clinical practice in these patients.

DETAILED DESCRIPTION:
This is a prospective cohort study that will enroll patients who are about to or have already undergone DBS electrode placement for a variety of disorders including, but not limited to Parkinson's disease, essential tremor, dystonia, depression, epilepsy, neuropathic pain and Alzheimer's disease. This eligible patient population is broad but unified by the fact that they will all undergo DBS to treat specific circuit dysfunctions. Pre-operative DBS patients and patients with externalized leads or internalized IPG may be included.

We propose to study patients with externalized leads or internalized IPG programmed at either 'switched off' (IPG at 0 volt and off state) and 'switched on' settings We have already performed phantom safety testing for these experimental conditions and found it to be safe. We propose to perform the following scans:

1. Structural 1.5Tesla or 3Tesla MRI with 8 channel coil/or transmit-receive head coil - 3D FSPGR, standard FRFSE T2 scan, standard DTI scan (white matter tracts) and standard QSM (Quantitative Susceptibility Mapping) scan (Iron quantification).
2. Resting state and task based functional MRI with 8 channel coil

Further, we propose to assess whether the aforementioned scans can be used as an adjunct to improve current DBS post-operative follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years of age
* Participants must be planned to undergo, or have undergone implantation of DBS electrodes
* Participants must be able to understand the purpose of this research and must sign the informed consent form.
* Participants must understand that the role of this research is to enhance our understanding of brain functioning and that he/she will not directly or indirectly benefit from the study.

Exclusion Criteria:

* Participants who have serious cognitive or psychological impairments and cannot give informed consent.
* Participants who are unable to effectively or efficiently communicate, for example patients suffering from speech deficits (dysarthria, aphasia) or are non-English speaking.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Brain areas engaged with deep brain stimulation | 3 months before DBS implant to 1 year after DBS implant.
  The primary outcome of interest is safety of 3T structural and functional brain MRI scans in patients with implanted DBS.

SECONDARY OUTCOMES:
Structural connectivity using 1.5T or 3T MRI | 3 months before DBS implant to 1 year after DBS implant.
  • to study volume changes (mm3) associated with DBS therapy in patients with movement disorders, psychiatric illness, epilepsy, and pain
Functional connectivity using 1.5T or 3T MRI | 3 months before DBS implant to 1 year after DBS implant.
  • To study the mechanisms underlying the therapeutic effects of DBS as measured by changes in functional and anatomical connectivity of the motor, sensory, memory and cognition circuits.
Clinical outcome | 3 months before DBS implant to 1 year after DBS implant.
  • number of clinic visits required until optimization

CONTACTS AND LOCATIONS:
Overall Officials: Andres Lozano, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boutet A, Madhavan R, Elias GJB, Joel SE, Gramer R, Ranjan M, Paramanandam V, Xu D, Germann J, Loh A, Kalia SK, Hodaie M, Li B, Prasad S, Coblentz A, Munhoz RP, Ashe J, Kucharczyk W, Fasano A, Lozano AM. Predicting optimal deep brain stimulation parameters for Parkinson's disease using functional MRI and machine learning. Nat Commun. 2021 May 24;12(1):3043. doi: 10.1038/s41467-021-23311-9. PMID 34031407